CLINICAL TRIAL: NCT05036876
Title: Insulin Degludec Versus Glargine U300 for the Management of Hospitalized Patients With Type 2 Diabetes: Randomized Controlled Trial
Brief Title: Degludec Glargine U300 Hospital Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medanta, The Medicity, India (Other)
Responsible Party: Principal Investigator, Dr Mohammad Shafi Kuchay, Senior Consultant, Medanta, The Medicity, India
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MMDHS01
Record Dates: First submitted 2021-08-27; First posted 2021-09-08 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-12

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — insulin degludec

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Degludec (Experimental): Study participants with type 2 diabetes undergoing elective coronary artery bypass graft (CABG) surgery will receive 100% of the total daily dose (TDD) given as a basal bolus regimen with degludec once daily plus rapid-acting insulin glulisine before meals.
  Degludec insulin 100 Units/mL, average dose: 30-40 U/day; Insulin glulisine 100 Units/mL, average dose: 20-40 U/day
  Interventions: Drug: Degludec
- Glargine U300 (Active Comparator): Study participants with type 2 diabetes undergoing CABG surgery will receive 100% of the total daily dose (TDD) given as a basal bolus regimen with glargine U300 once daily plus rapid-acting insulin glulisine before meals.
  Glargine U300;300 Units/mL, average dose: 30-40 U/day; Insulin glulisine 100 Units/mL, average dose: 20-40 U/day
  Interventions: Drug: Glargine U300

INTERVENTIONS:
Drug: Degludec — Treatment with insulin degludec when compared to insulin glargine U-300 will result in similar blood glucose control in hospitalized patients with type 2 diabetes.
  Arms: Degludec
Drug: Glargine U300 — Treatment with insulin glargine U300 when compared to insulin degludec will result in similar blood glucose control in hospitalized patients with type 2 diabetes.
  Arms: Glargine U300

SUMMARY:
Limited data exist about the use of insulin degludec and insulin glargine U300 in the hospitalized patients. A previous study compared the safety and efficacy of insulin degludec versus insulin glargine U100 for the management of hospitalized patients with type 2 diabetes. However, there is no data comparing the efficacy and safety of insulin degludec versus insulin glargine U300 for the management of hospitalized patients with type 2 diabetes. Accordingly, the proposed study will provide a clinically useful information on the efficacy (blood glucose control) and safety (hypoglycemia) of insulin degludec versus insulin glargine U300 for the management of hospitalized patients with type 2 diabetes.

DETAILED DESCRIPTION:
The purpose of this study is to find out if treatment with insulin degludec when compared to insulin glargine U300 will result in similar blood sugar control in hospitalized patients with type 2 diabetes.

Primary outcome measure

1. Change in mean daily blood glucose concentration in hospitalized patients [ Time Frame: The first 7 days of therapy ] Blood glucose will be measured before each meal, bedtime and at 3:00 am. Mean daily blood glucose concentration will be calculated to determine differences in inpatient glycemic control in patients with type 2 diabetes treated with basal bolus regimen or basal plus regimen with insulin degludec or glargine U300 once daily plus insulin glulisine before meals.

Secondary outcome measures

1. Number of basic glucose readings between 70 mg/dl and 180 mg/dl before meals in hospitalized patients.

   Blood glucose will be measured before each meal, bedtime and at 3:00 am, and proportion of basic glucose readings between 70 mg/dl and 180 mg/dl will be recorded.
2. Number of hypoglycemic episodes (BG < 70 mg/dl and 54 mg/dl) in hospitalized patients.

   Blood glucose will be measured before each meal, bedtime and 3:00 am, and number of hypoglycemic episodes (< 70 mg/dl and 54 mg/dl) will be recorded.
3. Number of severe hypoglycemia (< 54 mg/dl) episodes in hospitalized patients Blood glucose will be measured before each meal, bedtime and at 3:00 am, and number of hypoglycemia (< 54 mg/dl) episodes will be recorded.
4. Number of episodes of severe hyperglycemia (BG > 240 mg/dl) in hospitalized patients Blood glucose will be measured before each meal, bedtime and at 3:00 am, and number of severe hyperglycemia (> 240 mg/dl) episodes will be recorded.
5. Daily dose of basal insulin, daily dose of prandial insulin, and total daily dose in hospitalized patients The study team will document day and time of insulin administration of study drug given once daily and prandial- rapid-acting insulin (aspart) given before meals. The study team will also record dose and number of units given as supplement (correction) to correct hyperglycemia.
6. Average blood glucose (mg/dl), percentage time in target, percentage time below target, and percentage time above target in a subgroup of study participants A subgroup of participants (n = 100) will be monitored using continuous glucose monitoring system (CGMS) (FreeStyle Libre).

Eligibility criteria

Inclusion Criteria:

1. Males or females >30 years admitted to the hospital for elective CABG surgery.
2. A known history of T2D treated either with diet alone, oral monotherapy, any combination of oral antidiabetic agents, short-acting GLP1-RA (exenatide, liraglutide) or insulin therapy except for degludec and glargine U300.
3. Study participants must have a randomization total daily dose (TDD) insulin requirement of at least 20 units per day.
4. Signed, informed consent prior to any study procedures.

Exclusion Criteria:

1. Subjects with increased BG concentration, but without a known history of diabetes (stress hyperglycemia).
2. Subjects treated with diet alone (no antidiabetic agents) and admission HbA1c <7%.
3. Subjects with a history of diabetic ketoacidosis and hyperosmolar hyperglycemic state, or ketonuria.
4. Patients treated with degludec or glargine U300, or with long-acting weekly GLP1-RA (weekly exenatide, dulaglutide or albiglutide).
5. Patients with history of clinically relevant hepatic disease (diagnosed liver cirrhosis and portal hypertension), ongoing corticosteroid therapy (equal to a prednisone dose ≥5 mg/day), or impaired renal function (eGFR< 30 ml/min), or congestive heart failure (NYHA- IV).
6. Patients with medical and surgical pancreatic disease.
7. Mental condition rendering the subject unable to understand the nature, scope, and possible consequences of the study.
8. Known or suspected allergy to trial medication(s), excipients, or related products.

Sample size calculation

Noninferiority for the primary end point of glycemic control was defined as a mean blood glucose difference of <18 mg/dL between degludec and glargine U300. A blood glucose difference of such a magnitude has been reported in other superiority trials as nonclinically significant and is smaller than significant treatment effects. Assuming the true blood glucose difference between the treatment groups is zero, and using one-sided, two-sample t tests, we required 90 subjects for each treatment group to achieve 90% power. Accounting for a 10% attrition rate, we aimed to enrol 220 subjects in total to achieve >90% power.

Interventions Experimental: Degludec Study participants with type 2 diabetes undergoing coronary artery bypass graft (CABG) surgery will receive 100% of the total daily dose (TDD) given as a basal bolus regimen with degludec once daily plus rapid-acting insulin glulisine before meals.

Degludec insulin 100 Units/mL, average dose: 30-40 U/day. Insulin Glulisine, 100 Units/mL, average dose: 20-40 U/day.

Drug: Degludec Degludec is a long-acting human insulin analog indicated to improve glycemic control in adults with diabetes mellitus. Patients will be treated with bolus regimen given half of total daily dose (TDD) as basal once daily and half as glulisine divided in three equal doses before meals. Patients with poor oral intake or with medical instruction to withhold oral intake (NPO) will receive the basal dose, but prandial dose will be held. Insulin dose will be adjusted daily to maintain a fasting and pre-dinner BG between 100 mg/dl and 180 mg/dl.

Drug: Rapid-acting insulin Rapid-acting insulin will be given in three equally divided doses before each meal. To prevent hypoglycemia, if a subject is not able to eat, aspart insulin dose will be held.

Active Comparator: Glargine U300

Study participants with type 2 diabetes undergoing CABG surgery will receive 100% of the total daily dose (TDD) given as basal bolus regimen with glargine U300 once daily plus rapid-acting insulin glulisine before meals.

Insulin glargine (U300), 300 Units/mL, average dose: 30-40 U/day. Rapid-acting insulin glulisine, 100 Units/mL, average dose: 20-40 U/day.

Drug: Glargine (U300)

Glargine U300 is a long-acting human insulin analog indicated to improve glycemic control in adults with diabetes mellitus. Patients will be treated with bolus regimen given half of total daily dose (TDD) as basal once daily and half as insulin glulisine divided in three equal doses before meals. Patients with poor oral intake or with medical instruction to withhold oral intake (NPO) will receive the basal dose, but prandial dose will be held. Insulin dose will be adjusted daily to maintain a fasting and pre-dinner BG between 100 mg/dl and 180 mg/dl.

Drug: Rapid-acting insulin glulisine Glulisine insulin will be given in three equally divided doses before each meal. To prevent hypoglycemia, if a subject is not able to eat, glulisine insulin dose will be held.

Glucose monitoring Glucose levels will be assessed by capillary point-of-care (POC) testing before meals, bedtime and at 3:00 am.

A subgroup of participants (n = 100) will be monitored with a professional (blinded) Abbott FreeStyle Libre continuous glucose monitoring (CGM).

ELIGIBILITY:
Inclusion Criteria:

1. Males or females 30 years or above admitted to the hospital for elective CABG surgery
2. A known history of type 2 diabetes treated with any combination of oral antidiabetic agents, short-acting GLP1-RA (exenatide, liraglutide) or insulin therapy except for degludec and glargine U300.
3. Study participants must have a randomization total daily dose (TDD) insulin requirement of at least 20 units per day.
4. Signed, informed consent prior to any study procedures.

Exclusion Criteria:

1. Subjects with increased BG concentration, but without a known history of diabetes (stress hyperglycemia).
2. Subjects treated with diet alone (no antidiabetic agents) and admission HbA1c <7%.
3. Subjects with a history of diabetic ketoacidosis and hyperosmolar hyperglycemic state, or ketonuria.
4. Patients treated with degludec or glargine U300, or with long-acting weekly GLP1-RA (weekly exenatide, or dulaglutide).
5. Patients with history of clinically relevant hepatic disease (diagnosed liver cirrhosis and portal hypertension), ongoing corticosteroid therapy (equal to a prednisone dose ≥5 mg/day), or impaired renal function (eGFR< 30 ml/min), or congestive heart failure (NYHA- IV).
6. Patients with medical and surgical pancreatic disease.
7. Mental condition rendering the subject unable to understand the nature, scope, and possible consequences of the study.
8. Known or suspected allergy to trial medication(s), excipients, or related products.

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Actual)
Dates: Start 2021-10-10 (Actual); Primary Completion 2022-03-01 (Actual); Study Completion 2022-03-01 (Actual)

PRIMARY OUTCOMES:
Change in mean daily blood glucose concentration in hospitalized patients | The first 7 days of therapy
  Blood glucose will be measured before each meal, bedtime and at 3:00 am. Mean daily blood glucose concentration will be calculated to determine differences in inpatient glycemic control in patients with type 2 diabetes treated with basal bolus regimen or basal plus regimen with insulin degludec or glargine U-300 once daily plus aspart insulin before meals.

SECONDARY OUTCOMES:
Number of basic glucose readings between 70 mg/dl and 180 mg/dl before meals in hospitalized patients | The first 7 days of therapy
  Blood glucose will be measured before each meal, bedtime and at 3:00 am, and proportion of basic glucose readings between 70 mg/dl and 180 mg/dl will be recorded.
Number of hypoglycemic episodes (BG < 70 mg/dl and 54 mg/dl) in hospitalized patients | The first 7 days of therapy
  Blood glucose will be measured before each meal, bedtime and 3:00 am, and number of hypoglycemic episodes (< 70 mg/dl and 54 mg/dl) will be recorded
Number of severe hypoglycemia (< 54 mg/dl) episodes in hospitalized patients | The first 7 days of therapy
  Blood glucose will be measured before each meal, bedtime and at 3:00 am, and number of hypoglycemia (< 54 mg/dl) episodes will be recorded
Number of episodes of severe hyperglycemia (BG > 240 mg/dl) in hospitalized patients | The first 7 days of therapy
  Blood glucose will be measured before each meal, bedtime and at 3:00 am, and number of severe hyperglycemia (> 240 mg/dl) episodes will be recorded
Daily dose of basal insulin, daily dose of prandial insulin, and total daily dose in hospitalized patients | The first 7 days of therapy
  The study team will document day and time of insulin administration of study drug given once daily and prandial- rapid-acting insulin (aspart) given before meals. The study team will also record dose and number of units given as supplement (correction) to correct hyperglycemia
Average blood glucose (mg/dL), percentage time in target, percentage time below target, and percentage time above target in a subgroup of study participants. | The first 7 days of therapy
  A subgroup of participants (n = 100) will be monitored using continuous glucose monitoring system (CGMS) (FreeStyle Libre).

CONTACTS AND LOCATIONS:
Locations (1):
- Division Of Endocrinology and Diabetes , Medanta The Medicity Hospital, Gurgaon, Haryana, India

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared after a reasonable request
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code

REFERENCES:
- [Result] Umpierrez GE, Hor T, Smiley D, Temponi A, Umpierrez D, Ceron M, Munoz C, Newton C, Peng L, Baldwin D. Comparison of inpatient insulin regimens with detemir plus aspart versus neutral protamine hagedorn plus regular in medical patients with type 2 diabetes. J Clin Endocrinol Metab. 2009 Feb;94(2):564-9. doi: 10.1210/jc.2008-1441. Epub 2008 Nov 18. PMID 19017758
- [Result] Umpierrez GE, Smiley D, Jacobs S, Peng L, Temponi A, Mulligan P, Umpierrez D, Newton C, Olson D, Rizzo M. Randomized study of basal-bolus insulin therapy in the inpatient management of patients with type 2 diabetes undergoing general surgery (RABBIT 2 surgery). Diabetes Care. 2011 Feb;34(2):256-61. doi: 10.2337/dc10-1407. Epub 2011 Jan 12. PMID 21228246
- [Result] Pasquel FJ, Gianchandani R, Rubin DJ, Dungan KM, Anzola I, Gomez PC, Peng L, Hodish I, Bodnar T, Wesorick D, Balakrishnan V, Osei K, Umpierrez GE. Efficacy of sitagliptin for the hospital management of general medicine and surgery patients with type 2 diabetes (Sita-Hospital): a multicentre, prospective, open-label, non-inferiority randomised trial. Lancet Diabetes Endocrinol. 2017 Feb;5(2):125-133. doi: 10.1016/S2213-8587(16)30402-8. Epub 2016 Dec 8. PMID 27964837
- [Result] Umpierrez GE, Smiley D, Hermayer K, Khan A, Olson DE, Newton C, Jacobs S, Rizzo M, Peng L, Reyes D, Pinzon I, Fereira ME, Hunt V, Gore A, Toyoshima MT, Fonseca VA. Randomized study comparing a Basal-bolus with a basal plus correction insulin regimen for the hospital management of medical and surgical patients with type 2 diabetes: basal plus trial. Diabetes Care. 2013 Aug;36(8):2169-74. doi: 10.2337/dc12-1988. Epub 2013 Feb 22. PMID 23435159